CLINICAL TRIAL: NCT00883363
Title: Reduction of Myocardial Infarction by Preconditioning in Patients With Ruptured Abdominal Aortic Aneurysm
Acronym: PreconRAAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nikolaj Eldrup (Other)
Collaborators: Aarhus University Hospital (Other); Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor-Investigator, Nikolaj Eldrup, MD PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NE_RAAA_PRECON_01
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: precondition; ruptured abdominal aortic aneurysm; myocardial infarction
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precondition (Experimental): Induction of precondition at start of operation on a arm
  Interventions: Procedure: Precondition
- Control (No Intervention): No precondition

INTERVENTIONS:
Procedure: Precondition — Precondition on a arm in four intervals at start of surgery for ruptured aortic aneurysm
  Arms: Precondition

SUMMARY:
Preconditioning in patients treated for elective abdominal aneurysm showed that the rate of perioperative myocardial infarction could be reduced by 80 %(ARR from 27% to 5%). Precondition where performed by 10 minutes of clamping of each iliac arteries before clamping the abdominal aorta. Human studies in cardiac patients have shown promising results with precondition. Instead of clamping arteries they have all performed the procedure by inflating a blood pressure cuff above arterial pressure on a arm.

The investigators want to investigate if preconditioning induced by a blood pressure cuff on a arm can reduce the perioperative rate of myocardial infarction in patients open operated for ruptured abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ruptured abdominal aortic aneurysm offered surgery
* Age > 18 years

Exclusion Criteria:

* Technical inoperable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in myocardial infarction | 4 to 5 years

SECONDARY OUTCOMES:
Improvement in survival Description on inflammatory response | 4 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Eldrup, MD PhD, Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus university hospital skejby department of cardio thoracic and vascular surgery, Aarhus, Region Midt, Denmark

REFERENCES:
- [Derived] Pedersen TF, Budtz-Lilly J, Petersen CN, Hyldgaard J, Schmidt JO, Kroijer R, Gronholdt ML, Eldrup N. Randomized clinical trial of remote ischaemic preconditioning versus no preconditioning in the prevention of perioperative myocardial infarction during open surgery for ruptured abdominal aortic aneurysm. BJS Open. 2018 Mar 26;2(3):112-118. doi: 10.1002/bjs5.55. eCollection 2018 Jun. PMID 29951634
- See also: Study homepage with information — http://web.me.com/eldrup/forsk/